CLINICAL TRIAL: NCT04817449
Title: Molecular Spectroscopy in Identification and Assessment of Ovarian Cancer
Brief Title: Spectroscopy in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-21-12
Record Dates: First submitted 2021-03-04; First posted 2021-03-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms; Ovary Cyst; Ovary Disease
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Cysts; Ovarian Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Histological sections of tissue specimens of ovary, omentum or peritoneum Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected Ovarian Cancer: Patients referred or self presenting to secondary care with signs or symptoms of ovarian cancer.

SUMMARY:
Ovarian cancer is the eighth most common cause of cancer death in the world. Advanced stage at diagnosis is associated with lower survival rates, thus early detection appears to have an important role.

Raman Spectroscopy is a non-invasive technique that uses the interaction of light to identify the composition of the sample tested.

The aim of the project is to explore the use of spectroscopic techniques in the detection of ovarian cancer. There are two different assessments within the project:

1. Identify ovarian cancer in blood - Raman spectroscopic analysis will be performed on blood plasma taken from patients with suspected ovarian cancer.
2. Detect active cancer within post chemotherapy fibrotic tissue - Ex vivo Raman spectroscopic analysis of peritoneal, omental or ovarian tissues collected from patients undergoing surgical treatment for ovarian cancer.

The results of the spectroscopy will be correlated to clinical outcome and histological diagnosis respectively.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Symptoms suggestive of ovarian cancer
* Patients undergoing treatment of Ovarian Cancer

Exclusion Criteria:

* Less than 18 years of age
* Unable to consent to the study due to communication difficulties
* Unable to consent to the study due to lack of capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to secondary care with suspected ovarian cancer symptoms. Patients with likely ovarian cancer, yet to start definitive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Ascertain the diagnostic performance of vibrational spectroscopy for detection of Ovarian Cancer | 2 years
  Biomarkers for ovarian cancer will be identified by analysing Raman spectral data of plasma samples taken from patient with ovarian cancer symptoms. Clinical outcome of cancer/no cancer will be used to correlate the results.
Ascertain the discriminatory ability of vibrational spectroscopy to differentiate between normal, fibrotic and cancerous tissue | 2 years
  Samples taken from post chemotherapy patients will be analysed to identify the spectral signature of ovarian cancer in chemotherapy exposed tissue.

SECONDARY OUTCOMES:
Performance of vibrational spectroscopy in chemotherapy response prediction | 2 years
  Plasma samples after 1st cycle of chemotherapy will be analysed to evaluate for changes in biomarkers after chemotherapy treatment.
Performance of vibrational spectroscopy in recurrence prediction | 2 years
  Plasma samples after recurrence of cancer will be analysed and compared to initial spectral signature at diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Bristol and Weston NHS Trust, Bristol, United Kingdom